CLINICAL TRIAL: NCT06260904
Title: Efficacy and Safety of add-on Apremilast Versus add-on Methotrexate in Patients With Oral Lichen Planus: A Randomized Controlled Trial
Brief Title: Efficacy and Safety of add-on Apremilast Versus add-on Methotrexate in Patients With Oral Lichen Planus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, Dr. Monalisa Jena, M.D., Additional Professor, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIIMS BBSR/PGThesis/23-24/112
Record Dates: First submitted 2024-01-25; First posted 2024-02-15 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Oral Lichen Planus
Keywords: Lichen planus; Oral lichen planus; Prednisolone; Methotrexate; Apremilast; IL 6; VAS; PGA
MeSH Terms: conditions — Lichen Planus, Oral; Lichen Planus | interventions — Prednisolone; apremilast; Methotrexate

STUDY DESIGN:
Intervention Model Description: randomized, add-on, active-controlled, open-label, parallel-design clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prednisolone and Methotrexate (Control Arm) (Active Comparator): prednisolone 0.75mg/kg/day (a maximum dose of 30mg at baseline) and Methotrexate 15 mg weekly for 12 weeks.
  Interventions: Drug: Prednisolone; Drug: Methotrexate
- Prednisolone and Apremilast (Test Arm) (Experimental): prednisolone 0.75mg/kg/day (a maximum dose of 30mg at baseline) and Apremilast 30 mg twice daily for 12 weeks.
  Interventions: Drug: Prednisolone; Drug: Apremilast

INTERVENTIONS:
Drug: Prednisolone — prednisolone 0.75mg/kg/day (a maximum dose of 30mg at baseline) orally
Drug: Apremilast — Apremilast 30 mg twice daily orally
  Arms: Prednisolone and Apremilast (Test Arm)
Drug: Methotrexate — Methotrexate 15 mg weekly orally
  Arms: Prednisolone and Methotrexate (Control Arm)

SUMMARY:
Lichen planus is an inflammatory disorder of unknown aetiology affecting the stratified squamous epithelia, with an estimated global prevalence of 0.22 to 0.5 %. Oral mucosa (Oral Lichen Planus; OLP) is the most commonly affected region. Corticosteroids are the primary treatment of choice. A prolonged treatment with steroids is required for clinical improvement, which increases the chances of long-term adverse effects. So, there is a need for newer, effective treatment modalities, such as retinoids, methotrexate, Janus kinase inhibitors, PDE4 inhibitors, etc.

Of these, methotrexate is a dihydrofolate reductase inhibitor that inhibits the replication and function of T and B lymphocytes. It has shown a good response to OLP (around 83%) in a study by Lajevardi et al. and can be considered a treatment option in patients with moderate to severe OLP. Apremilast is a drug with a novel immunomodulatory mechanism of action. It inhibits phosphodiesterase type IV, which increases levels of cyclic adenosine monophosphate (cAMP), thus activating protein kinase A and inhibiting various inflammatory mediators. Based on a pilot study by Paul et al., apremilast is associated with clinical improvement in lichen planus.

Among the various treatment options, there is a lack of head-on trials. Methotrexate is an immunosuppressant with various systemic adverse effects and requires close monitoring. Whereas apremilast is a non-immunosuppressive drug with a better safety profile, it does not show such adverse effects. These drugs can be used as an add-on to low-dose steroids in view of reducing the adverse effects associated with steroid therapy. To the best of our knowledge, there is no randomized controlled trial comparing these two drugs to date. Hence, the present study has been planned to evaluate the safety and efficacy of methotrexate versus apremilast as an add-on to the standard steroid therapy in OLP patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 of either sex with the clinical diagnosis of oral lichen planus.
* Patients with a PGA score of ≥3 (moderate and severe oral LP).
* Patient not responding to topical or intralesional corticosteroid.
* Patients who are willing to give informed written consent.

Exclusion Criteria:

* Treatment with a systemic corticosteroid within the last 4 weeks.
* Patients on any immunosuppressive agents such as azathioprine, cyclosporine and others within one month of recruitment.
* Patients with clinical history and any lesion distribution suspicious of a lichenoid drug eruption and patients with other skin diseases.
* Past or current history of any malignancy including moderate to severe dysplasia of the oral mucosa on oral biopsy.
* Severe active infection, including active tuberculosis, hepatitis B or C infection
* Patients with cytopenia (Hb <9g/dl, leukocyte count <4000/mm3, platelet count <100,000/mm3)
* Patient with history of alcohol abuse.
* Decreased liver or renal function (creatinine > 2.0mg/dl, total bilirubin > 2.5 mg/dl).
* Severe acute infection, uncontrolled diabetes mellitus, untreated glaucoma, congenital or acquired immunodeficiency, active gastroduodenal ulcer, severe osteoporosis, severe cardiac disease (NYHA grade IV), MI in the last four weeks, severe schizophrenia or depression.
* Patient with a history of hypersensitivity to Methotrexate or Apremilast.
* Pregnancy and lactation, women of childbearing age without effective contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-01-26 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Pain by Visual Analogue Scale (VAS) score | 8 weeks and 12 weeks
  Change in Visual Analogue Scale (VAS) score after treatment with prednisolone and methotraxate Vs Prednisolone and Apremilast at baseline, 8 weeks and 12 weeks. The VAS consists of a 10 cm line, with two endpoints representing 0 ('no pain') and 10 ('pain as bad as it could possibly be') interpretation of the scores: 0 =No Pain 2 = Mild 4 = Nagging 6 =Miserable 8 =Intense 10 = Worst

SECONDARY OUTCOMES:
Severity by Physician global assessment of disease (PGA) score | 8 weeks and 12 weeks
  compare the proportion of patients achieving a reduction of Physician global assessment of disease (PGA) score of 0 or a 2-grade reduction (minimum initial PGA 3) after treatment with prednisolone and methotraxate Vs Prednisolone and Apremilast at baseline, 8 weeks and 12 weeks by using a 6-point disease severity scoring system.
  (0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe, 5=very severe).
Severity and pain by oral mucosal disease severity score | 8 weeks and 12 weeks
  the change in oral mucosal disease severity score (maximum 106) after treatment with prednisolone and methotraxate Vs Prednisolone and Apremilast at baseline, 8 weeks and 12 weeks.
  Total score = Site score + Activity score + pain Score (Maximum 106) higher scores indicating greater disease activity
serum IL 6 level | 12 weeks
  Change in serum IL 6 after treatment with prednisolone and methotraxate Vs Prednisolone and Apremilast he levels of salivary and serum IL-6 were significantly higher among patients with OLP than among healthy control participants
Quality of life by using oral health-related quality of life score (ORAL HEALTH IMPACT PROFILE - 14 ) | 8 weeks and 12 weeks
  Change in the oral health-related quality of life from baseline after 8 and 12 weeks.
  designed to assess patients' perception of the impact of oral disorders on their quality of life (QoL).
  The OHIP-14 scores can range from 0 to 56 and are calculated by summing the ordinal values for the 14 items. The domain scores can range from 0 to 8. Higher OHIP-14 scores indicate worse and lower scores indicate better OHRQol
Incidence of treatment-emergent adverse events of both test and control group | 12 weeks
  treatment-emergent adverse events in both the groups The adverse events in the patients are to be assessed by non-directive questioning at the time of the follow-up visit. Patients can access the investigators directly in case of any adverse events and report them. All adverse events irrespective of their previous reported status are to be recorded with details about nature, intensity, duration, measures taken, outcome, and causal relationship to prednisolone, methotrexate and apremilast.

CONTACTS AND LOCATIONS:
Overall Officials: Debasish Hota, MD, DM, Study Director — Professor
Locations (1):
- AIIMS Bhubaneswar, Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gorouhi F, Davari P, Fazel N. Cutaneous and mucosal lichen planus: a comprehensive review of clinical subtypes, risk factors, diagnosis, and prognosis. ScientificWorldJournal. 2014 Jan 30;2014:742826. doi: 10.1155/2014/742826. eCollection 2014. PMID 24672362
- [Background] Farhi D, Dupin N. Pathophysiology, etiologic factors, and clinical management of oral lichen planus, part I: facts and controversies. Clin Dermatol. 2010 Jan-Feb;28(1):100-8. doi: 10.1016/j.clindermatol.2009.03.004. PMID 20082959
- [Background] Solimani F, Forchhammer S, Schloegl A, Ghoreschi K, Meier K. Lichen planus - a clinical guide. J Dtsch Dermatol Ges. 2021 Jun;19(6):864-882. doi: 10.1111/ddg.14565. Epub 2021 Jun 7. PMID 34096678
- [Background] Veneri F, Bardellini E, Amadori F, Conti G, Majorana A. Efficacy of ozonized water for the treatment of erosive oral lichen planus: a randomized controlled study. Med Oral Patol Oral Cir Bucal. 2020 Sep 1;25(5):e675-e682. doi: 10.4317/medoral.23693. PMID 32683383
- [Background] Le Cleach L, Chosidow O. Clinical practice. Lichen planus. N Engl J Med. 2012 Feb 23;366(8):723-32. doi: 10.1056/NEJMcp1103641. No abstract available. PMID 22356325
- [Background] Mohan RPS, Gupta A, Kamarthi N, Malik S, Goel S, Gupta S. Incidence of Oral Lichen Planus in Perimenopausal Women: A Cross-sectional Study in Western Uttar Pradesh Population. J Midlife Health. 2017 Apr-Jun;8(2):70-74. doi: 10.4103/jmh.JMH_34_17. PMID 28706407
- [Background] Kanwar AJ, De D. Methotrexate for treatment of lichen planus: old drug, new indication. J Eur Acad Dermatol Venereol. 2013 Mar;27(3):e410-3. doi: 10.1111/j.1468-3083.2012.04654.x. Epub 2012 Jul 24. PMID 22827806
- [Background] Lajevardi V, Ghodsi SZ, Hallaji Z, Shafiei Z, Aghazadeh N, Akbari Z. Treatment of erosive oral lichen planus with methotrexate. J Dtsch Dermatol Ges. 2016 Mar;14(3):286-93. doi: 10.1111/ddg.12636. PMID 26972194
- [Background] Chauhan P, De D, Handa S, Narang T, Saikia UN. A prospective observational study to compare efficacy of topical triamcinolone acetonide 0.1% oral paste, oral methotrexate, and a combination of topical triamcinolone acetonide 0.1% and oral methotrexate in moderate to severe oral lichen planus. Dermatol Ther. 2018 Jan;31(1). doi: 10.1111/dth.12563. Epub 2017 Nov 10. PMID 29124831
- [Background] Papp K, Reich K, Leonardi CL, Kircik L, Chimenti S, Langley RG, Hu C, Stevens RM, Day RM, Gordon KB, Korman NJ, Griffiths CE. Apremilast, an oral phosphodiesterase 4 (PDE4) inhibitor, in patients with moderate to severe plaque psoriasis: Results of a phase III, randomized, controlled trial (Efficacy and Safety Trial Evaluating the Effects of Apremilast in Psoriasis [ESTEEM] 1). J Am Acad Dermatol. 2015 Jul;73(1):37-49. doi: 10.1016/j.jaad.2015.03.049. PMID 26089047